CLINICAL TRIAL: NCT02076113
Title: Cervical Spondylotic Myelopathy Surgical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCID: 2013-085; CE-1304-6173 (Other: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cervical Spondylosis With Myelopathy
Keywords: cervical spondylotic myelopathy; degenerative cervical spondylosis; spinal fusion
MeSH Terms: interventions — Decompression; Gene Fusion; Laminoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ventral (Active Comparator): Ventral Decompression with Fusion
  Interventions: Procedure: Ventral (Front) decompression with Fusion
- Dorsal (Active Comparator): Dorsal Decompression with Fusion or Dorsal Laminoplasty
  Interventions: Procedure: Dorsal (Back) Decompression with Fusion; Procedure: Dorsal (back) Laminoplasty

INTERVENTIONS:
Procedure: Ventral (Front) decompression with Fusion — Ventral decompression and fusion will be performed using a multi-level discectomy (including partial or single level corpectomy) with fusion and plating. Allograft will be used at each disc space and all compressive osteophytes will be removed using the operating microscope. Fixation will be performed with rigid, semi-constrained, or dynamic titanium plates to optimize fusion and minimize complications.
  Other Names: Anterior Cervical Discectomy and Fusion (ACDF)
  Arms: Ventral
Procedure: Dorsal (Back) Decompression with Fusion — Dorsal decompression and fusion will be performed using midline cervical laminectomy with the application of lateral mass screws and rods for rigid fixation. All surgeons will use local bone and allograft as needed to perform a lateral mass fusion, which typically will include one level rostral to the levels decompressed.
  Other Names: Posterior decompression and fusion
  Arms: Dorsal
Procedure: Dorsal (back) Laminoplasty — Laminoplasty will be performed using an open-door approach with the application of plates and screws at each treated level. Ceramic or allograft laminar spacers (surgeon's choice) can be used with plates and screws to expand the canal diameter.
  Arms: Dorsal

SUMMARY:
The purpose of the study is to determine the optimal surgical approach (ventral vs dorsal) for patients with multi-level cervical spondylotic myelopathy (CSM). There are no established guidelines for the management of patients with CSM, which represents the most common cause of spinal cord injury and dysfunction in the US and in the world.

This study aims to test the hypothesis that ventral surgery is associated with superior Short Form-36 physical component Score (SF-36 PCS) outcome at one year follow-up compared to dorsal approaches and that both ventral and dorsal surgery improve symptoms of spinal cord dysfunction measured using the modified Japanese Orthopedic Association Score (mJOA). A secondary hypothesis is that health resource utilization for ventral surgery, dorsal fusion, and laminoplasty surgery are different. A third hypothesis is that cervical sagittal balance post-operatively is a significant predictor of SF-36 PCS outcome.

DETAILED DESCRIPTION:
Patients' images will be transmitted electronically (without identifying information) to a group of 15 CSM surgeon investigators for their expert opinion. They will provide their opinion on surgical strategy. Equipoise for randomization will be established using this spinal experts network polling mechanism.

If randomized, the patient will be randomized to one of the two treatment approaches - either Ventral (front) (treatment A) or Dorsal (back) (treatment B) approach. If randomized to treatment A (front surgery), the patient will receive decompression/fusion from the front of the neck. If randomized to treatment B (dorsal/back surgery), then the patient and their surgeon will select which posterior procedure they will receive (either dorsal decompression/fusion or dorsal laminoplasty).

Treatment A: Decompression/fusion from the front of the neck.

Treatment B: Dorsal/posterior neck surgery (one of the two surgical procedures listed below):

Dorsal decompression/fusion or dorsal laminoplasty (no fusion)

Functional outcomes will be determined using well-known quantitative scales (SF-36, Oswestry Neck Disability Index (NDI), mJOA, and EuroQol-5D). These instruments will be administered pre-op, 3 months, 6 months, and at 1 year. Additionally, functional outcomes instruments (SF-36, Oswestry Neck Disability Index, and EuroQol-5D) will be collected annually at years 2,3,4 and 5.

Pre-op imaging will include a cervical MRI and cervical CT as well as cervical flexion/extension films and standing cervical-thoracic-lumbar-sacral x-ray . A cervical MRI will be performed at 3 months. At 1 year (randomized patients only) will undergo cervical flexion/ extension xrays and standing cervical-thoracic-lumbar-sacral x-ray . A cervical CT will be performed only if the Oswestry NDI score is > 30.

ELIGIBILITY:
Inclusion Criteria:

* CSM (≥2 levels of spinal cord compression from C3 to C7)
* Present with ≥2 of the following symptoms/signs: clumsy hands, gait disturbance, hyperreflexia, up going toes, bladder dysfunction.

Exclusion Criteria:

* C2-C7 kyphosis>5º (measured in standing neutral cervical spine radiograph),
* Segmental kyphotic deformity (defined by ≥3 osteophytes extending dorsal to a C2-C7 dorsal-caudal line measured on cervical spine CT),
* Structurally significant ossification of posterior longitudinal ligament (OPLL - measured on cervical spine CT),
* Previous cervical spine surgery
* Significant active health-related co-morbidity (Anesthesia Class IV or higher).

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2025-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Ghogawala, MD, Principal Investigator — Lahey Clinic, Inc.
Locations (16):
- United States (15):
  - University of California- San Francisco, San Francisco, California
  - Emory, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Washington University School of Medicine- St. Louis, St Louis, Missouri
  - Rutgers-New Jersey Medical School, Newark, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Columbia, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MetroHealth, Cleveland, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah Health Sciences, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University Health Network-University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available after publication of the trial's primary outcome results. Requests can be emailed to zoher.ghogawala@lahey.org.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after publication of the trial's primary results.
Access Criteria: Researchers whose proposed use of data has been approved with a signed data use agreement.

REFERENCES:
- [Background] Ghogawala Z, Martin B, Benzel EC, Dziura J, Magge SN, Abbed KM, Bisson EF, Shahid J, Coumans JV, Choudhri TF, Steinmetz MP, Krishnaney AA, King JT Jr, Butler WE, Barker FG 2nd, Heary RF. Comparative effectiveness of ventral vs dorsal surgery for cervical spondylotic myelopathy. Neurosurgery. 2011 Mar;68(3):622-30; discussion 630-1. doi: 10.1227/NEU.0b013e31820777cf. PMID 21164373
- [Background] Ghogawala Z, Coumans JV, Benzel EC, Stabile LM, Barker FG 2nd. Ventral versus dorsal decompression for cervical spondylotic myelopathy: surgeons' assessment of eligibility for randomization in a proposed randomized controlled trial: results of a survey of the Cervical Spine Research Society. Spine (Phila Pa 1976). 2007 Feb 15;32(4):429-36. doi: 10.1097/01.brs.0000255068.94058.8a. PMID 17304133
- [Background] Ghogawala Z, Benzel EC, Heary RF, Riew KD, Albert TJ, Butler WE, Barker FG 2nd, Heller JG, McCormick PC, Whitmore RG, Freund KM, Schwartz JS. Cervical spondylotic myelopathy surgical trial: randomized, controlled trial design and rationale. Neurosurgery. 2014 Oct;75(4):334-46. doi: 10.1227/NEU.0000000000000479. PMID 24991714
- [Background] Roguski M, Benzel EC, Curran JN, Magge SN, Bisson EF, Krishnaney AA, Steinmetz MP, Butler WE, Heary RF, Ghogawala Z. Postoperative cervical sagittal imbalance negatively affects outcomes after surgery for cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2014 Dec 1;39(25):2070-7. doi: 10.1097/BRS.0000000000000641. PMID 25419682
- [Background] Ghogawala Z, Terrin N, Dunbar MR, Breeze JL, Freund KM, Kanter AS, Mummaneni PV, Bisson EF, Barker FG 2nd, Schwartz JS, Harrop JS, Magge SN, Heary RF, Fehlings MG, Albert TJ, Arnold PM, Riew KD, Steinmetz MP, Wang MC, Whitmore RG, Heller JG, Benzel EC. Effect of Ventral vs Dorsal Spinal Surgery on Patient-Reported Physical Functioning in Patients With Cervical Spondylotic Myelopathy: A Randomized Clinical Trial. JAMA. 2021 Mar 9;325(10):942-951. doi: 10.1001/jama.2021.1233. PMID 33687463
- [Derived] Miranda SP, Whitmore RG, Kanter A, Mummaneni PV, Bisson EF, Barker FG 2nd, Harrop J, Magge SN, Heary RF, Fehlings MG, Albert TJ, Arnold PM, Riew KD, Steinmetz MP, Wang MC, Heller JG, Benzel EC, Ghogawala Z. Patients May Return to Work Sooner After Laminoplasty: Occupational Outcomes of the Cervical Spondylotic Myelopathy Surgical Trial. Neurosurgery. 2025 Jan 1;96(1):131-141. doi: 10.1227/neu.0000000000003048. Epub 2024 Jun 24. PMID 38912784
- See also: Patient Centered Outcomes Research Institute — https://www.pcori.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between April 1, 2014 and March 30, 2018 from 15 study sites.
Pre-assignment Details: 269 participants were eligible and enrolled; 163 randomized for treatment and 91 enrolled in a non-randomized cohort because either 80% or greater of review panel selected one surgical approach over the other (76), the participant did not consent to randomization (13), or at least 50% of review panel did not favor randomization (equipoise). 15 withdrew prior to randomization. Primary analysis compared ventral surgical approach to dorsal surgical approach.
Period: Overall Study
Arm/Group | Ventral | Dorsal
Started | 63 | 100
Surgery as Randomized | 62 (1 patient underwent dorsal fusion surgery) | 96 (4 patients underwent ventral fusion surgery)
3-Month Follow-up | 56 (5 missed follow-up visit; 2 lost to follow-up) | 90 (9 missed follow-up appointment; 1 lost to follow-up)
6-Month Follow-up | 53 (7 missed follow-up visit; 3 lost to follow-up) | 91 (7 missed follow-up visit; 1 lost to follow-up; 1 deceased)
1-Year Follow-up | 60 (3 lost to follow-up) | 95 (2 missed follow-up visit; 1 lost to follow-up; 2 deceased)
2-Year Follow-up | 51 (5 missed follow-up visit; 4 lost to follow-up; 2 withdrew consent; 1 deceased) | 79 (14 missed follow-up visit; 1 lost to follow-up; 3 withdrew consent; 3 deceased)
Completed | 56 | 93
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Death | 1 | 3

BASELINE CHARACTERISTICS:
Population: Primary analysis compared ventral surgical approach to dorsal surgical approach for treatment of cervical spondylotic myelopathy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ventral | Dorsal | Total
Number analyzed (Participants) | 63 | 100 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (7.2) | 62.5 (8.8) | 62.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 51 | 80
  Male | 34 | 49 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 61 | 96 | 157
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 54 | 85 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 5 | 10
  United States | 58 | 95 | 153
Baseline work status [Count of Participants; unit: Participants] — Population: 63/63 ventral participants and 98/100 dorsal participants reported their baseline work status.
  Participants
    number analyzed (Participants) | 63 | 98 | 161
    Working full-time | 17 | 40 | 57
    Retired | 14 | 29 | 43
    Not working, unable to work | 17 | 18 | 35
    Not working but able to work | 8 | 7 | 15
    Working part-time | 7 | 4 | 11
ASA physical status class [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) physical status classification is used to assess a patient's physical health and comorbidities to predict perioperative risk prior to surgery. Patients with class IV status (systemic disease that is life threatening) or higher were excluded from the study. Population: 61/63 ventral participants and 98/100 dorsal participants have reported ASA physical status class.
  Participants
    number analyzed (Participants) | 61 | 98 | 159
    1 (healthy) | 0 | 1 | 1
    II (mild systemic disease) | 31 | 46 | 77
    III (significant systemic disease) | 30 | 51 | 81
Number of stenotic levels [Mean (Standard Deviation); unit: levels] — Stenosis is the narrowing of the spinal canal, which causes the spinal cord to be compressed. The number of stenotic levels are the number of affected levels in the cervical spine that are causing the compression on the spinal cord and may contribute to the signs and symptoms the patient presents with.
  levels | 2.8 (0.7) | 2.8 (0.8) | 2.8 (0.7)
Number of stenotic levels [Count of Participants; unit: Participants] — Stenosis is the narrowing of the spinal canal, which causes the spinal cord to be compressed. The cervical vertebrae between C2 and T1 were included in the CSM-S trial. Patients presented with 1 to 5 levels of stenosis.
  Participants
    1 | 0 | 3 | 3
    2 | 22 | 29 | 51
    3 | 33 | 55 | 88
    4 | 8 | 11 | 19
    5 | 0 | 2 | 2
Neck Disability Index (NDI) score [Mean (Standard Deviation); unit: units on a scale] — The Neck Disability Index (NDI) ranges from 0 to 100, with lower scores representing less disability. A typical patient with moderate neck pain and disability would have a score between 20 and 40.
  units on a scale | 38.6 (19.1) | 35.3 (20.4) | 36.6 (19.9)
SF-36 mental component score [Mean (Standard Deviation); unit: units on a scale] — Short Form 36 (SF-36) mental component summary score ranges from 0 to 100, with higher scores representing better quality of life. A typical patient with cervical myelopathy who is being recommended surgery would have a score between 30 and 40.
  units on a scale | 45.6 (12.2) | 46.6 (12.1) | 46.2 (12.1)
SF-36 physical component score [Mean (Standard Deviation); unit: units on a scale] — Short Form 36 (SF-36) physical component summary (PCS) score ranges from 0 to 100, with higher scores representing better quality of life. A typical patient with cervical myelopathy who is being recommended surgery would have a score between 30 and 40.
  units on a scale | 37.4 (8.8) | 37.3 (9.9) | 37.3 (9.5)
mJOA scale score [Mean (Standard Deviation); unit: units on a scale] — The modified Japanese Orthopedic Association (mJOA) scale ranges from 0 to 17, with higher scores representing less dysfunction due to myelopathy. A typical patient with moderate cervical myelopathy has an mJOA score between 12 and 14. Many surgical studies show that patients with cervical myelopathy have mJOA scores in this range.
  units on a scale | 12.2 (2.7) | 12.1 (2.2) | 12.2 (2.4)
EQ-5D score [Mean (Standard Deviation); unit: units on a scale] — For the Euro-Qol 5 Dimensions (EQ-5D) score, 0 indicates death and 1 indicates a perfect health state. EQ-5D scores between 0.6 and 0.7 represent a moderate but significant reduction in the overall health-related quality of life.
  units on a scale | 0.64 (0.21) | 0.61 (0.21) | 0.62 (0.21)
EQ-5D visual analog scale score [Mean (Standard Deviation); unit: units on a scale] — For the EQ-5D visual analog scale, patients scores their health state on a scale from 0 to 100, with higher scores representing better health.
  units on a scale | 61.7 (20.9) | 63.1 (21.7) | 62.5 (21.3)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Change in Short Form 36 (SF 36) Physical Component Score (PCS) From Baseline to 1 Year and 2 Year
Description: Standardized measure of patient's functional health and well being as reported by the patient. The SF-36 physical component summary (PCS) scores range from 0 to 100, with higher scores representing better quality of life.
Time Frame: 1 year and 2 year
Population: Primary analysis was conducted as-randomized (ventral vs. dorsal). At 1 year, there were 60/63 ventral participants and 95/100 dorsal participants available for analysis. At 2 year, there were 51/63 ventral participants and 79/100 dorsal participants available for analysis. Estimated mean change was calculated from the baseline SF-36 PCS score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ventral | Dorsal
Number analyzed (Participants) | 60 | 97
units on a scale
  1 year: number analyzed (Participants) | 60 | 95
  1 year | 5.9 (8.2) | 6.2 (10.2)
  2 year: number analyzed (Participants) | 51 | 79
  2 year | 5.2 (7.9) | 6.0 (11.0)

2. Secondary Outcome: Short Form-36 (SF-36) Physical Component Summary (PCS) Score
Description: Standardized measure of patient's functional health and well being as reported by the patient. The SF-36 physical component summary (PCS) scores range from 0 to 100, with higher scores representing better quality of life. A typical patient with cervical myelopathy who is being recommended surgery would have a score between 30 and 40.
Time Frame: Pre-operative, 1 year and 2 year
Population: Secondary outcomes in the primary analysis were analyzed as-randomized (ventral vs. dorsal). At 1 year, there were 60/63 ventral participants and 95/100 dorsal participants available for analysis. At 2 year, there were 51/63 ventral participants and 79/100 dorsal participants available for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ventral | Dorsal
Number analyzed (Participants) | 60 | 97
units on a scale
  Pre-operative | 37.6 (8.9) | 37.6 (9.9)
  1 year: number analyzed (Participants) | 60 | 95
  1 year | 43.5 (10.7) | 44.0 (10.5)
  2 year: number analyzed (Participants) | 51 | 79
  2 year | 43.4 (10.5) | 43.6 (10.8)

3. Secondary Outcome: Oswestry Neck Disability Index (NDI)
Description: Standard instrument for measuring self-rated disability secondary to neck pain. The NDI ranges from 0 to 100, with lower scores representing less disability. A typical patient with moderate neck pain and disability would have a score between 20 and 40.
Time Frame: Pre-operative, 1 year and 2 year
Population: Secondary outcomes in the primary analysis were analyzed as-randomized (ventral vs. dorsal). At 1 year, there were 60/63 ventral participants and 97/100 dorsal participants available for analysis. At 2 year, there were 51/63 ventral participants and 79/100 dorsal participants available for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ventral | Dorsal
Number analyzed (Participants) | 60 | 97
units on a scale
  Pre-operative | 38.1 (19.1) | 35.4 (20.5)
  1 year: number analyzed (Participants) | 60 | 95
  1 year | 22.9 (20.1) | 22.5 (20.3)
  2 year: number analyzed (Participants) | 51 | 79
  2 year | 20.4 (20.2) | 22.1 (21.3)

4. Secondary Outcome: EuroQol-5D
Description: Standardized measure of health related quality of life. For the EQ-5D score, 0 indicates death and 1 indicates a perfect health state. EQ-5D scores between 0.6 and 0.7 represent a moderate but significant reduction in overall health-related quality of life.
Time Frame: Pre-operative, 1 year and 2 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ventral | Dorsal
Number analyzed (Participants) | 60 | 97
units on a scale
  Pre-operative | 0.64 (0.21) | 0.61 (0.21)
  1 year: number analyzed (Participants) | 59 | 95
  1 year | 0.77 (0.21) | 0.76 (0.19)
  2 year: number analyzed (Participants) | 51 | 79
  2 year | 0.78 (0.20) | 0.78 (0.19)

5. Secondary Outcome: Modified Japanese Orthopedic Association Score mJOA
Description: Short instrument for the functional assessment of patients. The scale ranges from 0 to 17, with higher scores representing less dysfunction due to myelopathy. A typical patient with moderate cervical myelopathy has an mJOA score between 12 and 14.
Time Frame: Pre-operative and 1 year
Population: Secondary outcomes in the primary analysis were analyzed as-randomized (ventral vs. dorsal). At 1 year, there were 60/63 ventral participants and 91/100 dorsal participants available for analysis. At 2 year, there were 51/63 ventral participants and 79/100 dorsal participants available for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ventral | Dorsal
Number analyzed (Participants) | 60 | 91
units on a scale
  Pre-operative | 12.2 (2.7) | 12.2 (2.3)
  1 year | 14.5 (2.6) | 14.2 (2.5)

6. Secondary Outcome: Sagittal Balance Measurements
Description: Sagittal vertical axis was measured at 1 year postoperatively.
Time Frame: 1 year
Population: Secondary outcomes in the primary analysis were analyzed as-randomized (ventral vs. dorsal). At 1 year, there were 49/63 ventral participants and 78/100 dorsal participants available for analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ventral | Dorsal
Number analyzed (Participants) | 49 | 78
mm | 23.2 (11.8) | 26.7 (13.3)

7. Secondary Outcome: Cumulative Health Resource Utilization Over 1 Year by Actual Treatment Groups - Ventral Fusion, Dorsal Fusion, and Dorsal Laminoplasty
Description: Patient diary capturing out of pocket health utilization related to cervical surgery. The cumulative health resource utilization over 1-year is reported for the 'as treated' cohorts. Patients reported diagnostic imaging (MRI, x-ray, or CT), along with physical therapy and ongoing (at 1 year) physical therapy, opioid use and ongoing (at 1 year) opioid use, along with appointments with physicians. Data was collected at 1, 3, and 6 months and 1 year after surgery. The data presented is accumulative over the 1 year after surgery.
Time Frame: Within 1 year of surgery
Population: All patients reported diagnostic imaging (MRI, x-ray, or CT), along with physical therapy and ongoing (at 1 year) physical therapy, opioid use and ongoing (at 1 year) opioid use, along with appointments with physicians. Data was collected at 1, 3, and 6 months after surgery, as well as at 1 year. The data presented is accumulative over the 1 year after surgery.
Measure: Number; unit: occurrences
Groups:
- Dorsal Decompression With Fusion: Dorsal (Back) Decompression with Fusion: Dorsal decompression and fusion will be performed using midline cervical laminectomy with the application of lateral mass screws and rods for rigid fixation. All surgeons will use local bone and allograft as needed to perform a lateral mass fusion, which typically will include one level rostral to the levels decompressed.
- Dorsal Laminoplasty: Dorsal (back) Laminoplasty: Laminoplasty will be performed using an open-door approach with the application of plates and screws at each treated level. Ceramic or allograft laminar spacers (surgeon's choice) can be used with plates and screws to expand the canal diameter.
Arm/Group | Ventral | Dorsal Decompression With Fusion | Dorsal Laminoplasty
Number analyzed (Participants) | 66 | 69 | 28
occurrences
  Diagnostic imaging | 52 | 60 | 17
  MRI | 28 | 32 | 11
  CT | 12 | 11 | 4
  x-ray | 50 | 51 | 13
  Physical Therapy | 34 | 39 | 13
  Ongoing physical therapy 1 year after surgery | 11 | 15 | 0
  Opioid use | 30 | 45 | 11
  Ongoing opioid use 1 year after surgery | 6 | 11 | 0
  Physician Appointments | 16 | 26 | 6

8. Secondary Outcome: Number of Participants With Continued Full or Part Time Work Status at Each Follow Up Time Point by Actual Treatment Groups - Ventral Fusion, Dorsal Fusion, and Dorsal Laminoplasty
Description: Work status was recorded for all patients (working full-time; working part-time; not working, unable to work; not working, but able to work; or retired) at each follow-up through 1 year.
Time Frame: Pre-operative, 1, 3 and 6 months and 1 year
Population: Only patients who were working either full- or part-time at baseline were included in the return to work analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ventral | Dorsal Decompression With Fusion | Dorsal Laminoplasty
Number analyzed (Participants) | 27 | 29 | 12
Participants
  Pre-operatively | 27 | 29 | 12
  1 month: number analyzed (Participants) | 25 | 28 | 11
  1 month | 9 | 5 | 6
  3 month: number analyzed (Participants) | 25 | 28 | 11
  3 month | 19 | 10 | 9
  6 month: number analyzed (Participants) | 24 | 26 | 11
  6 month | 19 | 16 | 8
  1 year: number analyzed (Participants) | 26 | 28 | 9
  1 year | 19 | 18 | 8

9. Secondary Outcome: Number of Participants With Complications by Actual Treatment Groups - Ventral Fusion, Dorsal Fusion, and Dorsal Laminoplasty
Description: Major complications included adverse events that were ongoing at 3 months, reoperations within 2 years, and 30-day readmissions. Minor complications were those that resolved within 3 months. All cases of postoperative motor radiculopathy were related to C5 nerve root dysfunction.
Time Frame: Complications were assessed at 2 years and categorized to have occurred within 30 days, 1 year or within 2 years.
Measure: Number; unit: participants
Arm/Group | Ventral | Dorsal Decompression With Fusion | Dorsal Laminoplasty
Number analyzed (Participants) | 66 | 69 | 28
participants
  Any Complications | 31 | 20 | 3
  Major complications | 14 | 15 | 2
  Prolonged dysphagia | 9 | 0 | 0
  Motor radiculopathy | 1 | 8 | 0
  Spinal cord injury | 0 | 0 | 1
  Deep vein thrombosis | 0 | 1 | 0
  Delayed wound healing | 0 | 1 | 0
  Minor complications | 18 | 5 | 1
  Dysphagia | 18 | 0 | 0
  Infection | 0 | 2 | 1
  Motor radiculopathy (resolved within 3 months) | 0 | 2 | 0
  Reoperations (within 2 year) | 4 | 4 | 0
  Readmissions (within 30 days) | 0 | 6 | 1
  Cervical (C5) paresis | 0 | 2 | 0
  Pulmonary embolism | 0 | 1 | 0
  Ileus | 0 | 1 | 0
  Uncontrolled neck pain | 0 | 1 | 0
  Infection (needing readmission) | 0 | 1 | 0
  Fever (unknown source) | 0 | 0 | 1

10. Secondary Outcome: Number of Participants With Unresolved Swallowing Difficulty (Complication) at 3 Months
Description: Dysphagia is considered swallowing difficulty. Difficulty swallowing that resolved within 3 months was considered a minor complication, while prolonged (on going after 3 months) dysphagia was considered a major complication.
Time Frame: 3 months, 1 year
Population: Complication were assessed by the actual treatment approach the participant received. 66 participants underwent ventral surgery and 97 participants underwent dorsal surgery.
Measure: Number; unit: participants
Arm/Group | Ventral | Dorsal
Number analyzed (Participants) | 66 | 69
participants
  Minor (resolved within 3 months) | 18 | 0
  Major (prolonged - ongoing after 3 month through 1 year follow-up) | 9 | 0

11. Other Pre Specified Outcome: Short Form-36 (SF-36) Physical Component Summary (PCS) Score by Actual Treatment Groups - Ventral Fusion, Dorsal Fusion, and Dorsal Laminoplasty
Description: Standardized measure of patient's functional health and well being as reported by the patient. The SF-36 physical component summary scores range from 0 to 100, with higher scores representing better quality of life.
Time Frame: Pre-operative, 1 year and 2 year
Population: At 1 year, 63/66 ventral participants, 66/69 dorsal decompression with fusion participants, and 26/28 dorsal laminoplasty participants were available for analysis. At 2 year, 54/66 ventral participants, 55/69 dorsal decompression with fusion participants, and 21/28 dorsal laminoplasty participants were available for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ventral | Dorsal Decompression With Fusion | Dorsal Laminoplasty
Number analyzed (Participants) | 63 | 68 | 26
units on a scale
  Pre-operative | 38.1 (9.1) | 37.3 (9.4) | 37.3 (11.1)
  1 year: number analyzed (Participants) | 63 | 66 | 26
  1 year | 43.8 (10.9) | 42.5 (10.4) | 47.1 (9.7)
  2 year: number analyzed (Participants) | 54 | 55 | 21
  2 year | 43.8 (10.7) | 41.5 (10.6) | 48.3 (9.3)

ADVERSE EVENTS:
Time Frame: Complications were assessed at 2 years and categorized to have occurred within 30 days, 1 year or within 2 years.
Description: Major complications included adverse events that were ongoing at 3 months, reoperations within 2 years, and 30-day readmissions. Minor complications were those that resolved within 3 months. All cases of postoperative motor radiculopathy were related to C5 nerve root dysfunction. Patients may have had more than 1 complication, so totals may be less that the sum of the categories.
Arm/Group | Ventral | Dorsal Decompression With Fusion | Dorsal Laminoplasty
All-Cause Mortality (participants affected / at risk) | 1/66 | 1/69 | 2/28
Serious Adverse Events (participants affected / at risk) | 14/66 | 15/69 | 2/28
Other Adverse Events (participants affected / at risk) | 18/66 | 5/69 | 1/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ventral (N=66) | Dorsal Decompression With Fusion (N=69) | Dorsal Laminoplasty (N=28)
Prolonged dysphagia (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0
Motor radiculopathy (ongoing at 3 months) (Musculoskeletal and connective tissue disorders) | 1 | 8 | 0 — All cases of postoperative motor radiculopathy were related to C5 nerve root dysfunction.
Spinal cord injury (Nervous system disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Delayed wound healing (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Reoperations (Surgical and medical procedures) | 4 | 4 | 0 — Reoperations within 2 years of index surgery.
Cervical (C5) paresis (readmissions within 30 days) (Nervous system disorders) | 0 | 2 | 0
Pulmonary Embolism (readmissions within 30 days) (Vascular disorders) | 0 | 1 | 0
Ileus (readmissions within 30 days) (Gastrointestinal disorders) | 0 | 1 | 0
Uncontrolled neck pain (readmissions within 30 days) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Infection (readmissions within 30 days) (General disorders) | 0 | 1 | 0
Fever (readmissions within 30 days) (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ventral (N=66) | Dorsal Decompression With Fusion (N=69) | Dorsal Laminoplasty (N=28)
Dysphagia (Musculoskeletal and connective tissue disorders) | 18 | 0 | 0
Infection (General disorders) | 0 | 2 | 1
Motor radiculopathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Delayed wound healing (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: CSM-S Randomized Clinical Trial - Primary Outcome - SF-36 (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02076113/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Cost-Effectiveness Analysis Plan (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT02076113/Prot_SAP_001.pdf